CLINICAL TRIAL: NCT01478503
Title: Double-blind, Randomized, Placebo-controlled, Dose-escalating, Exploratory Study to Investigate the Pharmacokinetics, Safety and Tolerability of Multiple Doses of YM178 OCAS-M in Healthy Young Male and Female Subjects and Healthy Elderly Male and Female Subjects
Brief Title: To Evaluate the Blood and Urine Concentration and the Safety and Tolerability of Increasing Repeated Doses of Mirabegron (YM178) OCAS in Healthy Young and Elderly Males and Healthy Young and Elderly Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 178-CL-031
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Pharmacokinetics; Healthy Subjects
Keywords: Pharmacokinetics; Mirabegron; Phase 1; Dose-Escalation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm A (Experimental): mirabegron
  Interventions: Drug: mirabegron OCAS
- Treatment Arm B (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mirabegron OCAS — oral
  Other Names: YM178 OCAS
  Arms: Treatment Arm A
Drug: Placebo — oral
  Arms: Treatment Arm B

SUMMARY:
The study aimed to compare age and gender differences for increasing doses of mirabegron when given to healthy young and elderly males and healthy young and elderly females.

DETAILED DESCRIPTION:
Each subject will receive a single dose of mirabegron OCAS-M or placebo on Day 2, followed by multiple dosing (qd) for 10 days (Day 5-14).

Young subjects will be divided into 4 groups and elderly subjects into 2 groups. Dosage will be different among groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young subjects aged 18-55 years (inclusive)
* Healthy elderly subjects aged 65-80 years (inclusive)
* Body weight between 60.0 and 100.0 kg (male) or between 50.0 and 90.0 kg (female), and Body Mass Index between 18.0 and 30.0 kg/m2

Exclusion Criteria:

* Known or suspected hypersensitivity to β-adrenergic receptor agonists or any components of the formulation used
* Any of the liver function tests (i.e. ALT, AST and bilirubin) above the upper limit of normal at repeated measures
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic as judged by the medical investigator.
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, electrocardiogram (ECG) and clinical laboratory tests
* Subjects taking β blockers or β agonists
* Use of any prescribed or Over-the-counter (OTC) drugs (including vitamins, natural and herbal remedies, e.g. St. John's wort) in the 2 weeks prior to admission to the Clinical Unit, except for occasional use of paracetamol (up to 3 g/day)
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampicin) in the 3 months prior to admission to the Clinical Unit
* Donation of blood or blood products within 3 months prior to admission to the Clinical Unit
* Any use of drugs of abuse, or smoking of more than 10 cigarettes (or equivalent) or more than 21 units of alcohol per week within the 3 months prior to study
* Participation in any clinical study within 3 months or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2005-05; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of mirabegron assessed by plasma concentration | Pre-dose until 72 hours after dosing

SECONDARY OUTCOMES:
Monitoring of safety and tolerability through assessment of vital signs, Electrocardiogram (ECG), clinical safety laboratory and adverse events | Baseline until 72 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (2):
- Netherlands (2):
  - Kendle Nederland, Utrecht
  - Pharma Bio Research, Zuidlaren

REFERENCES:
- [Background] Krauwinkel W, van Dijk J, Schaddelee M, Eltink C, Meijer J, Strabach G, van Marle S, Kerbusch V, van Gelderen M. Pharmacokinetic properties of mirabegron, a beta3-adrenoceptor agonist: results from two phase I, randomized, multiple-dose studies in healthy young and elderly men and women. Clin Ther. 2012 Oct;34(10):2144-60. doi: 10.1016/j.clinthera.2012.09.010. PMID 23063375